CLINICAL TRIAL: NCT00059592
Title: Valacyclovir in Immunocompromised Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Susan Blaney, Professor, Pediatrics-Hema & Oncology, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H6644
Record Dates: First submitted 2003-04-29; First posted 2003-04-30 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Shingles; Bone Marrow Transplantation
MeSH Terms: conditions — Herpes Zoster | interventions — Valacyclovir

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Valacyclovir (Experimental): oral Valacyclovir three times a day for 5 to 10 days.
  Interventions: Drug: Valacyclovir

INTERVENTIONS:
Drug: Valacyclovir
  Other Names: Valtrex

SUMMARY:
Shingles is an infection commonly seen in children with a weakened immune system (immunocompromised children). The immune system can be weakened as a result of medications that patients receive for cancer or other serious illness or as a result of a bone marrow transplantation. Shingles in children with a weakened immune system may spread throughout the body and in some instances may be life-threatening. Acyclovir is a medication that is routinely used to treat immunocompromised children with shingles in order to prevent further spread of their shingles and to help them heal faster. Acyclovir is also given to bone marrow transplant patients to prevent reactivation of HSV infection.

Valacyclovir is a new drug that is metabolized (broken down in the body) to acyclovir. Valacyclovir is given by mouth and studies done in adults have shown it to be more effective than acyclovir given by mouth.

The purpose of this study is to

* study the pharmacology of this drug (how the body handles this drug),
* determine if oral Valacyclovir can be safely given to children with shingles, and
* determine the type of side effects that occur when oral Valacyclovir is given to immunocompromised children.

DETAILED DESCRIPTION:
Patients with shingles:

Patients with shingles will receive oral Valacyclovir three times a day for 5 to 10 days. For the first 24 hours of treatment, patients will be admitted to the hospital for close monitoring. If there are no problems after the first 24 hours then the patient may be discharged to take the medicine at home.

After discharge patients will be seen and examined in clinic daily for the first 5 days, then on day 7 and after that every other day until the shingles show evidence of healing. A final physical exam and blood tests occur on day 21.

A small amount of fluid will be taken from one of the shingles lesions using a very fine needle to verify the presence of the virus that causes shingles. This will be done before the first dose of Valacyclovir and 3 days later.

Blood tests (no more than 2 teaspoons) will be performed twice a week to monitor for toxic effects of the drug. Blood samples will be drawn to evaluate the pharmacology of this drug(how the body handles the drug). Nine blood samples (less than one teaspoon each) will be obtained over 24 hours during the first day of treatment. The total amount of blood to be drawn is 9 teaspoons (3 tablespoons).

For children that are toilet trained, urine will be collected for 12 hours at the start of the study. This urine will be used to evaluate kidney function, and the pharmacology of valacyclovir. If there are unacceptable side effects or if there is evidence that the disease is spreading, despite being on Valacyclovir for more than 48 hours, then you will be taken off the study and started on acyclovir by vein.

Patients Undergoing Bone Marrow Transplantation:

Patients undergoing a bone marrow transplant will receive a single dose of valacyclovir in place of their first scheduled dose of acyclovir. They will then receive acyclovir as outlined by their physician.

Blood samples will be drawn to evaluate the pharmacology (how the body handles the drug) of the study drug. Fifteen blood samples (less than one teaspoon each) will be obtained over 24 hours during the first day of treatment. The total amount of blood to be drawn is 9 teaspoons (3 tablespoons. The total amount of blood drawn for all blood work including routine blood tests as well as pharmacokinetics will not be greater than 5% of the patients total blood volume. This amount of blood loss is a safe amount even for small children

ELIGIBILITY:
Inclusion Criteria:

* Patients must be >/= 2 and </= 18 years old.
* Patients must have a life expectancy of > 8 weeks.
* Patients must be receiving chemotherapy or have been treated with bone marrow transplantation or chemotherapy for an underlying malignancy or medical condition in the past 12 months, or have an underlying immunodeficiency syndrome.
* Patients must have adequate hepatic function (bilirubin ≤ 1.5 mg/dl: SGPT < 3x normal) and adequate renal function (creatinine ≤ 1.2 mg/dl or creatinine clearance ≥ 60 ml/min/1.73 m2).
* Acute Zoster Infection: Patients must have acute herpes zoster defined as </= 3 days of rash, limited to 3 or less dermatomes, and no evidence of dissemination (organ involvement e.g. hepatitis, pneumonitis, encephalitis).
* Patients must be able to swallow pills or tolerate a suspension of the medication.
* Children must be able to retain liquids at the time of enrollment.
* Written informed consent will be obtained from all patients and/or their parents prior to enrollment.
* Bone Marrow Transplant Patients: Patients without acute zoster infection, but with positive HSV serology who will be treated with acyclovir prophylaxis during the pretransplant period are eligible.

Exclusion Criteria:

* Patients with evidence of disseminated VZV infection, as documented by dermatomal zoster at more than 3 dermatomes.
* Patients with history of VZV infection > 3 days.
* Patients in relapse, (Stratum I only), or unstable medical conditions due to underlying disease.
* Patients with suspected acyclovir-resistant VZV infection.
* Patients who received systemic antiherpetic therapy in the previous 2 weeks before the onset of VZV infection.
* Patients with known history of adverse reaction to acyclovir in the past.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 1998-04-07 (Actual); Primary Completion 2004-12-30 (Actual); Study Completion 2005-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Blaney, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas